CLINICAL TRIAL: NCT00128414
Title: Treatment and Prevention of Pericarditis With Colchicine. A Multicenter Double Blind Randomized Trial. The CORP Trial: COlchicine for Recurrent Pericarditis
Brief Title: Study of Colchicine to Treat and Prevent Recurrent Pericarditis (First Episode)
Acronym: CORP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Sanitaria Locale 3, Torino (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCASL30501-2; EUDRACT number 2005-001570-28
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Pericarditis; Recurrence
Keywords: Pericarditis; Recurrence; Therapeutics; Prevention; Colchicine
MeSH Terms: conditions — Pericarditis; Recurrence | interventions — Colchicine; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo
- Colchicine (Experimental): Colchicine 1.0 mg twice daily for the first day followed by a maintenance dose of 0.5 mg twice daily for 6 month in patients ≥70 kg, and halved doses for patients <70 kg or intolerant to the highest dose.
  Interventions: Drug: Colchicine (for 6 months)

INTERVENTIONS:
Drug: Colchicine (for 6 months) — colchicine 1.0 mg twice daily for the first day followed by a maintenance dose of 0.5 mg twice daily for 1 month in patients ≥70 kg, and halved doses for patients <70 kg or intolerant to the highest dose.
  Arms: Colchicine
Drug: Placebo — Tablets identical in colour, shape, and taste were provided in blister packs.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether colchicine is safe and effective in the treatment and prevention of recurrent pericarditis (first episode).

DETAILED DESCRIPTION:
Colchicine is safe and effective in the management of recurrent pericarditis after failure of conventional treatment. Preliminary data have shown that it may be effective also in treatment of the first attack of recurrent pericarditis and the prevention of further recurrences.

Comparisons: The study will compare the safety and efficacy of colchicine in the treatment of the first attack of recurrent pericarditis and the secondary prevention of recurrences. Colchicine will be used in addition to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the first attack of recurrent pericarditis
* Age≥ 18 years
* Informed consent

Exclusion Criteria:

* Suspected neoplastic, tuberculous, or purulent etiology
* Known severe liver disease and/or elevated transaminases >1.5 times the upper limit of normality
* Serum creatinine >2.5 mg/dl
* Serum creatine kinase (CK) over the upper limit of normality or known myopathy
* Known gastrointestinal or blood disease
* Pregnant or lactating women or women not protected by a contraception method
* Known hypersensibility to colchicine
* Treatment with colchicine at enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 18 months

SECONDARY OUTCOMES:
Symptom persistence at 72 hours, remission rate at 1 week
Number of recurrences
Time to recurrence
Disease-related hospitalization, cardiac tamponade, constrictive pericarditis within the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rita TRINCHERO, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL 3 Torino; Massimo Imazio, MD, Study Chair — Cardiology Department. Maria Vittoria Hospital. ASL3 Torino.; Massimo Imazio, MD, Principal Investigator — Cardiology Department. Maria Vittoria Hospital. ASL3 Torino.
Locations (5):
- Italy (5):
  - Internal Medicine Dpt. Ospedali Riuniti, Bergamo, Bergamo
  - Department of Cardiology, San Maurizio Regional Hospital, Bolzano, Bolzano
  - Cardiology Dpt. Ospedale SS Annunziata, Savigliano, CN
  - Cardiology Department. Maria Vittoria Hospital. ASL3 Torino, Torino, Torino
  - Ospedale di Rivoli, Rivoli

REFERENCES:
- [Background] Imazio M, Cecchi E, Ierna S, Trinchero R; CORP Investigators. CORP (COlchicine for Recurrent Pericarditis) and CORP-2 trials--two randomized placebo-controlled trials evaluating the clinical benefits of colchicine as adjunct to conventional therapy in the treatment and prevention of recurrent pericarditis: study design and rationale. J Cardiovasc Med (Hagerstown). 2007 Oct;8(10):830-4. doi: 10.2459/JCM.0b013e3280110616. PMID 17885522
- [Derived] Imazio M, Brucato A, Cemin R, Ferrua S, Belli R, Maestroni S, Trinchero R, Spodick DH, Adler Y; CORP (COlchicine for Recurrent Pericarditis) Investigators. Colchicine for recurrent pericarditis (CORP): a randomized trial. Ann Intern Med. 2011 Oct 4;155(7):409-14. doi: 10.7326/0003-4819-155-7-201110040-00359. Epub 2011 Aug 28. PMID 21873705